CLINICAL TRIAL: NCT05465642
Title: Alterations of Gut Microbiota and Serum Biochemical Markers in Asian Patients With Drug-induced Liver Injury
Brief Title: Alterations of Gut Microbiota and Serum Biochemical Markers in DILI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Huikuan Chu, MD, Associate chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: UHCT22354
Record Dates: First submitted 2022-07-06; First posted 2022-07-20 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Drug-induced Liver Injury; Gut Microbiota; Biochemical Markers
Keywords: DILI; gut microbiota; serum biochemical markers
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — Retain patient blood and stool and extract DNA for identification of gut microbiota.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug-induced liver injury: history of taking hepatotoxic drugs, liver injury.
  Interventions: Other: Collect stool and blood samples from patients
- Healthy control: no liver disease or other disease
  Interventions: Other: Collect stool and blood samples from patients

INTERVENTIONS:
Other: Collect stool and blood samples from patients — Collect stool and blood samples from patients

SUMMARY:
Drug-induced liver injury is a leading cause of acute liver failure worldwide and one of the least understood areas in hepatology research. Increasing evidence has shown that drug-induced liver injury is associated with gut microbiota.

DETAILED DESCRIPTION:
Background:

Drug-induced liver injury(DILI) refers to the liver injury induced by all kinds of drugs and is the leading cause of acute liver failure worldwide. China has a large population base and a wide variety of clinical drugs, and it is common for the population to use drugs irregularly. Therefore, the incidence of DILI is increasing year by year. The pathogenesis of DILI is complicated, and there are often multiple mechanisms successively or altogether. As a result of the same effect, it is particularly important to study the pathogenesis of DILI and find its therapeutic target. Increasing evidence shows that DILI is related to the gut microbiota, which provides broader insights and opportunities for understanding and treating this disease.

Aims:

We aim to map the alterations of gut microbiota and serum biochemical markers in patients with DILI, and to investigate the effects and mechanisms of key strains on the development of DILI, providing a theoretical basis and potential targets for its treatment.

Methods:

Patients who meet the inclusion criteria will sign informed consent, their demographic data, clinical labs, serum, and feces will be collected at baseline. Fecal samples will be subject to 16S rRNA amplicon sequencing. Serum samples were taken for metabolomics detection.

Anticipated Results:

Compared to the healthy control group, patients with DILI will suffer from gut microbiota dysbiosis and have more microbes and microbial genes associated with inflammation and injury. The levels of serum biochemical markers are associated with the severity of DILI.

Implications and Future Studies:

Results of altered gut microbiome and serum biochemical markers could provide potential targets for manipulating intestinal microbiota to prevent or treat DILI.

ELIGIBILITY:
Inclusion Criteria:

1. The group of DILI:

1. aged >18 years;
2. patients who meet the diagnostic criteria of DILI in Guidelines for Diagnosis and Treatment of Drug-induced Liver Injury;
3. history of taking hepatotoxic drugs;
4. with relatively complete clinical data and good compliance.

2. The group of healthy control:

1. aged >18 years;
2. no history of liver disease and other diseases.

Exclusion Criteria:

1. with hepatocellular carcinoma (HCC) or hepatic metastases;
2. combined with infectious liver diseases, such as hepatitis A virus, hepatitis B virus, hepatitis C virus, hepatitis D virus, hepatitis E virus, and human immunodeficiency virus (HIV);
3. combined with non-infectious liver diseases, such as non-alcoholic fatty liver disease, alcoholic liver disease, autoimmune liver disease, immunoglobulin G4-related liver disease, Wilson's disease, alpha 1-antitrypsin deficiency, Budd-Chiari syndrome, and other congenital liver diseases;
4. combined with severe organic lesions of other organs;
5. pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy control will be recruited mainly from the outpatient or inpatient departments of Wuhan Union Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The changes of gut microbiota in the levels of phylum, genus, and species in two groups | 2 years
  The changes will be detected by genome sequencing
The different levels of serum aspartate transaminase/alanine transaminase (AST/ALT) in two groups | 2 years
  The changes will be detected by biochemical analyzers
The different levels of proinflammatory cytokines in two groups | 2 years
  The changes will be determined by ELISA kits
The changes of lncRNA and miRNA in two groups | 2 years
  The changes will be measured by quantitative polymerase chain reaction (qPCR)

CONTACTS AND LOCATIONS:
Overall Officials: Huikuan Chu, M.D., Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, wuhan
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Hartmann P, Chu H, Duan Y, Schnabl B. Gut microbiota in liver disease: too much is harmful, nothing at all is not helpful either. Am J Physiol Gastrointest Liver Physiol. 2019 May 1;316(5):G563-G573. doi: 10.1152/ajpgi.00370.2018. Epub 2019 Feb 15. PMID 30767680
- [Result] Wu G, Win S, Than TA, Chen P, Kaplowitz N. Gut Microbiota and Liver Injury (I)-Acute Liver Injury. Adv Exp Med Biol. 2020;1238:23-37. doi: 10.1007/978-981-15-2385-4_3. PMID 32323178
- [Result] Gong S, Lan T, Zeng L, Luo H, Yang X, Li N, Chen X, Liu Z, Li R, Win S, Liu S, Zhou H, Schnabl B, Jiang Y, Kaplowitz N, Chen P. Gut microbiota mediates diurnal variation of acetaminophen induced acute liver injury in mice. J Hepatol. 2018 Jul;69(1):51-59. doi: 10.1016/j.jhep.2018.02.024. Epub 2018 Mar 8. PMID 29524531
- [Result] Schneider KM, Elfers C, Ghallab A, Schneider CV, Galvez EJC, Mohs A, Gui W, Candels LS, Wirtz TH, Zuehlke S, Spiteller M, Myllys M, Roulet A, Ouzerdine A, Lelouvier B, Kilic K, Liao L, Nier A, Latz E, Bergheim I, Thaiss CA, Hengstler JG, Strowig T, Trautwein C. Intestinal Dysbiosis Amplifies Acetaminophen-Induced Acute Liver Injury. Cell Mol Gastroenterol Hepatol. 2021;11(4):909-933. doi: 10.1016/j.jcmgh.2020.11.002. Epub 2020 Nov 12. PMID 33189892
- See also: This web provides information of Human Subjects Protection in this study — https://gcp.whuh.com/index.aspx

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05465642/Prot_SAP_ICF_000.pdf